CLINICAL TRIAL: NCT02330809
Title: Drinking Extra Water To Prevent or Decrease Headaches - A Feasibility Online Randomized Controlled Trial With Adult Participants
Brief Title: Drinking Extra Water for to Prevent or Decrease Headaches
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study investigator retired and study not funded
Sponsor: ThinkWell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ThinkWell-PLOT-01
Record Dates: First submitted 2014-12-30; First posted 2015-01-05 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Headache
Keywords: headache; hunger intensity; public led online trial; water intake
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Daily extra water intake 2L (Experimental): Timing of daily extra water intake intervention-A: extra water intake: 8 8oz glasses of water a day (2L) - 2 first thing in the morning before breakfast, 2 before midday or midday meal, 2 before afternoon meal and 2 before evening meal.
  Intervention-B: Drink extra water at anytime over 24 hours
  Interventions: Other: Daily extra water intake; Other: Timing of daily extra water intake
- Daily extra water intake 1L (Experimental): Timing of daily extra water intake Intervention-A: 4 8oz glasses of water a day (1L) - 1 first thing in the morning before breakfast, 1 before midday or midday meal, 1 before afternoon meal and 1 before evening meal.
  Intervention-B: Drink extra water at anytime over 24 hours
  Interventions: Other: Daily extra water intake; Other: Timing of daily extra water intake
- Daily extra water intake 500ml (Experimental): Timing of daily extra water intake Intervention-A: 2 8oz glasses of water a day (500ml) - each half an hour before a meals
  Intervention-B: Drink extra water at anytime over 24 hours
  Interventions: Other: Daily extra water intake; Other: Timing of daily extra water intake
- Daily extra water intake 120ml (Experimental): Timing of daily extra water intake Intervention-A: 1/2 a glass of water on waking (120ml). If you forget to drink your water first thing, do not drink it later in the day, just skip this day and drink ½ a glass the next day on waking.
  Intervention-B: Drink extra water at anytime over 24 hours
  Interventions: Other: Daily extra water intake; Other: Timing of daily extra water intake

INTERVENTIONS:
Other: Daily extra water intake — Amount of extra daily water intake to consume
Other: Timing of daily extra water intake — Intervention-A: Timing of daily extra water intake specified Intervention-B: at any time during 24 hour period

SUMMARY:
The purpose of this study is to find out if drinking extra water helps people prevent or relieve headaches and hunger and, if so, what volume of water is most effective and when is it best to drink it?

DETAILED DESCRIPTION:
If participants decide to participate in this trial, they will be asked to drink a specific amount of water at particular times of the day for 14 days. A computer will decide by chance the amount of water they will be asked to drink each day of the trial and the times at which to drink this.

There are different amounts and different times that people will be asked to drink water, this is so that the investigators can find out if there is an optimal volume of water to drink, and a best time to drink water to reduce headaches or hunger. The least amount of water the computer could ask participants to drink is half a glass (that is 4oz or 120ml). The largest volume of water the computer could ask participants to drink would be eight glasses of water a day (a total of 64oz or 2L) spread across the day (that is not all at once). Once the computer has assigned participants to a particular volume and times to drink water, these will remain the same for every day throughout the study.

Participants will be asked to provide some brief information about themselves at the beginning of the study (for example, age, sex, height and whether you exercise, smoke or not). During the study they will be asked to weigh themselves and record this, Their dietary habits and the amount they drink will be kept on a private and confidential page on the study website. They will be asked to fill in [2] confidential short surveys about how they feel and their views, one at the start and one at the end of the study.

ELIGIBILITY:
Inclusion Criteria

* Any adult (defined as someone aged 18 or above) for whom advice to drink extra water is not contraindicated.

Exclusion Criteria

General exclusions

* < 18 years of age
* No personal email address
* Pregnancy
* Ecstasy recreational drug use

Exclusions Health Conditions

* Impaired renal function
* Chronic bowel problems
* Low sodium levels
* Diabetes insipidus
* Schizophrenia or history of psychosis
* Anorexia or bulimia
* Congestive heart failure
* Current chemotherapy treatment

Exclusions Concurrent Medications

* Taking regular non-steroidal anti-inflammatory drugs
* Diuretics (e.g. thiazides, indapamide, loop diuretics), also called "water tablets"
* Anti-depressants: Selective serotonin re-uptake inhibitors (SSRIs), Tricyclic and tetracyclic antidepressants (TCAs),monoamine oxidase inhibitor (MAOIs)
* Anti-psychotics (e.g. haloperidol)
* Anti-convulsants (e.g. sodium valproate, carbamazepine)
* Cancer drugs (anti-neoplastic agents)

Implicit exclusions

* People without internet access
* People who cannot read
* People without the ability to understand the website and informed consent documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of headache frequency/intensity | Daily for 14 days
  Online participant reported visual analog scales

SECONDARY OUTCOMES:
Hunger | Daily for 14 days
  Online participant reported Visual analog scales
Mood Questionnaire | Daily for 14 days
  Mood will be measured online using happy, sad, neutral faces
Body mass index (BMI) | Baseline and day 14
  Participants will use an automated online BMI calculator
Wellbeing | Baseline and day 14
  Patient Reported Outcome Measurement Information System (PROMIS) will be used to measure patient-reported outcome (PRO) for answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Burls, MD, Principal Investigator — ThinkWell and City University London; Amy I Price, PhD, Study Director — University of Oxford
Locations (1):
- ThinkWell, Oxford, Oxfordshire, United Kingdom